CLINICAL TRIAL: NCT00002276
Title: Study of Bleeding Tendency, Platelet Function, and Pharmacokinetics of Azidothymidine (AZT) and Motrin (Ibuprofen) in HIV-Infected Hemophiliacs
Brief Title: The Effects of AZT and Ibuprofen on HIV-Infected Patients With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 044A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-06

CONDITIONS: HIV Infections; Hemophilia A
Keywords: Blood Platelets; Ibuprofen; Drug Interactions; Zidovudine; Hemophilia A
MeSH Terms: conditions — HIV Infections; Hemophilia A | interventions — Ibuprofen; Zidovudine

INTERVENTIONS:
Drug: Ibuprofen
Drug: Zidovudine

SUMMARY:
To determine if platelet dysfunction and/or pharmacologic drug interaction occurs in patients taking both AZT and ibuprofen, which might account for enhanced bleeding tendency.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Hemophilia.
* HIV-seropositivity confirmed by Western Blot.

Prior Medication:

Required:

- AZT for study patients.

Allowed:

- Ibuprofen.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

Hospitalization for opportunistic infection, bacterial infection or malignancy.

Concurrent Medication:

Excluded:

* AZT (for control group).
* Antibiotics or other medication for opportunistic infection, bacterial infection, or malignancy.

Patients with the following prior conditions are excluded:

Hospitalization for opportunistic infection, bacterial infection, or malignancy.

Required:

* Ibuprofen.
* AZT 1-2 gm daily (for study patient) or not taking AZT (for control).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Ragni MV, Miller BJ, Whalen R, Ptachcinski R. Bleeding tendency, platelet function, and pharmacokinetics of ibuprofen and zidovudine in HIV(+) hemophilic men. Am J Hematol. 1992 Jul;40(3):176-82. doi: 10.1002/ajh.2830400305. PMID 1609771